CLINICAL TRIAL: NCT01091571
Title: The Effects of Oral Dipyridamole Treatment on the Innate Immune Response During Human Endotoxemia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: P. Pickkers MD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2009/347
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-03

CONDITIONS: Endotoxemia
Keywords: Adenosine; Endotoxin; Innate Immunity; Dipyridamole
MeSH Terms: conditions — Endotoxemia | interventions — Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endotoxemia placebo (Placebo Comparator): Endotoxin combined with placebo
  Interventions: Drug: Placebo; Other: LPS
- Endotoxemia Dipyridamole (Experimental): Endotoxin combined with Dipyridamol treatment
  Interventions: Drug: Dipyridamole; Other: LPS

INTERVENTIONS:
Drug: Dipyridamole — Oral treatment with dipyridamole 200 mg twice daily during seven consecutive days
  Other Names: Persantin retard
  Arms: Endotoxemia Dipyridamole
Drug: Placebo — Placebo twice daily during seven consecutive days
  Arms: Endotoxemia placebo
Other: LPS — The LPS derived from E. coli O:113 2ng/kg iv will be injected in 1 minute at a dosage of 2 ng/kg body weight.
  Other Names: Human endotoxemia

SUMMARY:
During sepsis and septic shock the immune response can be overwhelming leading to excessive tissue damage, organ failure and death. Ideally, the inflammatory response is modulated leading to both adequate protection to invading pathogens as well as limitation of an exuberant immune response. In the last few years adenosine is proposed to have a central role in the modulation of inflammation. In unfavorable conditions such as hypoxia, ischemia or inflammation adenosine is quickly up-regulated; with concentrations up to tenfold in septic patients. Many animal studies have shown that adenosine is able to attenuate the inflammatory response and decrease mortality rates. Therefore, pharmacological elevation of the adenosine concentration is an potential target to attenuate inflammation and limit organ injury. Dipyridamole, an adenosine re-uptake inhibitor is able to increase the adenosine concentration and limit ischemia-reperfusion injury. In order to study the effects of dipyridamole on the inflammatory response we aim to use the so called human endotoxemia model. This model permits elucidation of key players in the immune response to a gram negative stimulus in vivo, therefore serving as a useful tool to investigate potential novel therapeutic strategies in a standardized setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 35 years
* Male
* Healthy

Exclusion Criteria:

* Use of any medication.
* History of allergic reaction to dipyridamole
* Bleeding disorder.
* Smoking.
* Previous spontaneous vagal collapse.
* History, signs or symptoms of cardiovascular disease.
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complex bundle branch block.
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90).
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50).
* Renal impairment (defined as plasma creatinin >120 μmol/l).
* Liver enzyme abnormalities or positive hepatitis serology.
* Positive HIV serology or any other obvious disease associated with immune deficiency.
* Febrile illness in the week before the LPS challenge.
* Participation in another drug trial or donation of blood 3 months prior to the planned LPS challenge.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Circulating cytokines | 24 hours after LPS administration
  TNFx, IL6, IL10, IL1RA

SECONDARY OUTCOMES:
Hemodynamics | 24 hours after LPS administration
  Continious heart rate and blood pressure measurement
Sensitivity to norepinephrine | 24 hrs after LPS administration
  Venous occlusion plethysmography
Endothelial-dependent and independent vasorelaxation | 24 hours after LPS administration
  Venous occlusion plethysmography
Markers of endothelial damage and circulating endothelial cells | 24 hrs after LPS administration
  circulating adhesion molecules (ICAM, VCAM, E-selectin, P-selectin) circulating endothelial cells
Urinary excretion of markers of renal injury | 24 hrs after LPS administration
  GSTAlpha1-1 and GSTPi1-1
Adenosine and related nucleotide concentrations | 24 hrs after LPS administration
Additional blood samples will be drawn for genetic testing and measurement of: mRNA and proteins part of the adenosine metabolism | 24 hours after LPS administration
Oxydative stress | 24 hours after LPS administration
  Thiols, neutrophilic burst, calcium release of neuthrophils, TBARS, Carbonyls, FRAP, Myeloperoxidase, catalase, Griess assay

CONTACTS AND LOCATIONS:
Overall Officials: Bart P Ramakers, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Ramakers BP, Riksen NP, Stal TH, Heemskerk S, van den Broek P, Peters WH, van der Hoeven JG, Smits P, Pickkers P. Dipyridamole augments the antiinflammatory response during human endotoxemia. Crit Care. 2011;15(6):R289. doi: 10.1186/cc10576. Epub 2011 Nov 30. PMID 22129171